CLINICAL TRIAL: NCT02115555
Title: Advancing Diabetes Management in Adolescents Using Health Information Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tamara S. Hannon, Associate Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-04, IRB00000219
Record Dates: First submitted 2014-03-17; First posted 2014-04-16 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes
Keywords: type 1; diabetes; adolescents; heath information technology
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HIT-aided approach (Experimental): Adolescents and their parents randomized to this arm will be oriented on a HIT system. The system transmits self monitoring blood glucose self monitoring blood glucose data to a secure web portal. The subject will receive messages from the HIT system on the meter based upon the Self Monitored Blood glucose tests.
  Interventions: Behavioral: HIT-aided approach
- Contracted conflict management system (Experimental): Adolescent-parent pairs will meet with a health educator to establish a behavioral contract that will set patient-centered self-management goals for the adolescent.
  Interventions: Behavioral: Contracted conflict management system
- HIT plus contracted conflict management (Experimental): Adolescents and their parents randomized to this arm will be oriented on a HIT system. The system transmits self monitoring blood glucose data to a secure web portal. The subject will receive messages from the HIT system on the meter based upon the tests. In addition, adolescent-parent pairs will meet with a health educator to establish a behavioral contract that will set patient-centered self-management goals for the adolescent. This arm combines arms 1 and 2.
  Interventions: Behavioral: HIT plus contracted conflict management

INTERVENTIONS:
Behavioral: HIT-aided approach — Subjects randomized to this approach will be using the HIT-aided monitor.
  Arms: HIT-aided approach
Behavioral: Contracted conflict management system — Subjects randomized to this arm will be using the behavioral contracted conflict management system.
  Arms: Contracted conflict management system
Behavioral: HIT plus contracted conflict management — Subjects randomized to this arm will use both the HIT-aided approach and the behavioral contract conflict management system.
  Arms: HIT plus contracted conflict management

SUMMARY:
The study will compare three treatment strategies to look at the best clinical outcomes.

The investigator hypothesizes that the combined approach of a health information technology program plus a conflict-management contract will lead to the best outcomes.

DETAILED DESCRIPTION:
This study will compare three strategies for enhancing adherence to diabetes care in our population. The study will look at which strategy results in the best short-term clinical outcomes for the population. Also, the study will look at patient satisfaction of contact with his/her health care team, quality of life, and family dynamics.

The three arms are:

1. HIT (health information technology) aided approach
2. Contracted conflict-management strategy
3. Combination of the HIT-aided approach and the contracted conflict management strategy

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed for at least 6 months
* At least one or more parent/guardian who agrees to participate

Exclusion Criteria:

* Other chronic diseases with the exception of well-controlled asthma or treated thyroid disease

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Glycemic Control using HBA1C | Baseline, 3 months, and 6 months
  Change in Glycemic Control

SECONDARY OUTCOMES:
Frequency of self monitoring blood glucose measurement | Baseline, 3 months, 6 months
  change in Self-monitoring blood glucose measurement
Quality of Life | Baseline and 6 months
  Change in Diabetes-specific quality of life measures will be measured by the Varney's Pediatric Quality of Life 3.0 Diabetes Module.
Family dynamics | Baseline and 6 months
  Change in family dynamics measured by the Cornell Parent Behavior Description Scale and the Helping for Health Inventory.
Treatment Adherence Behaviors | Once per month for 6 months
  Change in treatment adherence behaviors measured by the Self-Care Inventory with supplemental questions determined by the investigator.

OTHER OUTCOMES:
Satisfaction | 3 month and 6 month
  Patient and parent satisfaction with the intervention with questions determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Hannon, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Riley Children's Specialties, Carmel, Indiana
  - Riley Children's Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No
Data will be shared via presentation and publications.